CLINICAL TRIAL: NCT07199309
Title: Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of MAR001 on Postprandial Lipids in Patients With Elevated Triglycerides and Remnant Cholesterol
Brief Title: A Mechanistic Study of MAR001 in Adults With Elevated Triglycerides and Remnant Cholesterol
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Marea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAR-104
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Hypertriglyceridemia
Keywords: Remnant Cholesterol; MAR001; Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MAR001 Dose (Experimental): Subcutaneous Injection
  Interventions: Drug: MAR001
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MAR001 — Subcutaneous Injection
  Arms: MAR001 Dose
Drug: Placebo — Subcutaneous Injection
  Arms: Matching Placebo

SUMMARY:
The primary objective of the study is to determine the effect of MAR001 as compared to placebo on levels of the triglycerides (TG) in the postprandial state in adults with elevated TG.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide informed consent and comply with the intervention and all study assessments
* Two fasting TG collected at two separate, consecutive visits at least 7 days apart during the Screening period
* HbA1c ≥ 5.7% and ≤ 8.5%
* Stable diet for a minimum of 3 months prior to screening and with no plans to change diet through duration of study
* Stable drug regimen (appropriate if relevant) prior to screening visit and no planned changes during screening or trial participation

Exclusion Criteria:

* Acute or chronic liver disease
* Diabetes medications (other than metformin)
* History of type 1 diabetes mellitus or history of diabetic ketoacidosis
* Newly diagnosed T2DM
* Participants with known active hepatitis A, B, or C
* Participants who are known to have uncontrolled human immunodeficiency virus (HIV) infection
* Uncontrolled hypothyroidism
* Any condition that prevents the participant from complying with study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in TG area under the curve after a mixed meal | 12 weeks
Change from baseline in peak plasma TG concentration after a mixed meal | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in RC area under the curve after a mixed meal | 12 weeks
Change from baseline in peak plasma RC concentration after a mixed meal | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Marea Site 301, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Undecided